CLINICAL TRIAL: NCT01993771
Title: Monitoring of Anaesthetic Depth at Different Locations in the Cerebral Cortex Using Bispectral Bilateral System
Brief Title: Monitoring of Anaesthesic Depth in the Cerebral Cortex Using Bispectral Bilateral System.
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Juan Luis Fernández Candil, MD, Parc de Salut Mar
Other Study IDs: HOLOBIS
Record Dates: First submitted 2013-09-20; First posted 2013-11-25 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Breast Surgery
MeSH Terms: interventions — Surgical Procedures, Operative; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Males and females with alopecia: Males and females with alopecia scheduled for general anaesthesia.
  Interventions: Procedure: Surgery with general anaesthesia.; Procedure: Raw EEG

INTERVENTIONS:
Procedure: Surgery with general anaesthesia.
Procedure: Raw EEG

SUMMARY:
This is a prospective, observational study, aimed to establish changes of bispectral bilateral system in both cerebral hemispheres during a total intravenous anaesthesia during breast surgery in the woman. By placing two Bispectral bilateral sensors (BIS), one on both frontal lobes, and another on both parietal lobes, we wanted to evaluate differences between frontal and parietal areas, when the patient is awake and during the anaesthetic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years old.
* Scheduled for general anaesthesia.
* Agree to participate(signed inform consent).

Exclusion Criteria:

* Neurological disease.
* Cognitive impairment.
* Egg allergy.
* Severe disease or condition that could potentially interfere with interpretation of tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with alopecia scheduled for general anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Bilateral BIS values from frontal and parietal areas. | Bilateral BIS values will be taken at baseline, anaesthetic induction, endotracheal intubation, skin incision, mantenance of anaesthesia and in emergence from anaesthesia ( 3 hours as a maximum from baseline to emergence).

SECONDARY OUTCOMES:
EEG changes at LOC (loss of consciousness) and ROC (recovery of consciousness). | Changes will be evaluated at induction and emergence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain